CLINICAL TRIAL: NCT00223795
Title: Walking Aids in the Management of Obesity-Related Knee Osteoarthritis
Brief Title: Walking Aids in the Management of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: F3873-R
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2014-04-22 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Obesity; Osteoarthritis
Keywords: Cane; Gait; Obesity; Osteoarthritis; Walking Aids
MeSH Terms: conditions — Obesity; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single point cane (Active Comparator): People with knee osteoarthritis underwent gait analysis with a cane
  Interventions: Device: Single point cane
- No cane (No Intervention): Patients with knee osteoarthritis undergo gait analysis without a cane

INTERVENTIONS:
Device: Single point cane — Participants with symptomatic knee osteoarthritis will undergo gait evaluation with and without a single point cane.
  Other Names: Guardian offset handled cane with sure grip
  Arms: Single point cane

SUMMARY:
The purpose of this study is to assess whether the single point cane will relieve pain and disability in overweight or obese people with knee OA through altered joint biomechanics and what factors influence acceptance of cane use.

DETAILED DESCRIPTION:
Knee OA is an important cause of disability and falls in overweight or obese individuals and limits their attempts at exercise and subsequent weight loss. Walking aids such as canes have been recommended in the management of knee OA in order to decrease pain by reducing loading across the knee and to increase physical activity. Little information is available regarding the impact of walking aids on psychosocial function and quality of life in individuals with limited mobility. No randomized controlled trials have studied the efficacy of walking aids on quality of life, pain, and function in overweight or obese individuals with symptomatic knee OA (5,6). The proposed research will evaluate the effects of walking aids in knee OA by testing the following hypothesis that the use of a single-point cane ipsilateral and contralateral to the affected limb will decrease pain from knee OA by altering gait biomechanics and will improve walking function and quality of life in overweight or obese individuals with symptomatic knee OA.

ELIGIBILITY:
Inclusion Criteria:

* 45-85 years old
* Able to walk 30 feet without postural sway and able to stand unaided
* Knee pain on movement with a WOMAC pain subscale of >35mm
* Documented osteoarthritis based on clinical and radiographic criteria
* Body Mass Index (BMI) > 25.0 - 29.9
* Ability to understand verbal and written instructions
* Ability to give informed consent determined by assessment of cognitive status

Exclusion Criteria:

* Concurrent medical/arthritic disease that could confound or interfere with evaluation of pain or efficacy. History of knee trauma or surgery, including arthroscopic surgery, in the past six months
* Severe obesity (weight > 300lbs)
* Upper body weakness
* Injury or amputation of the lower extremity joints
* History of other types of arthritis
* Spine, foot, or hip pain of sufficient magnitude to interfere with the evaluation of the index joint.
* Isolated patellofemoral disease manifested by primarily anterior knee pain in the absence of tibiofemoral radiographic finding.
* History of significant collateral or anterior cruciate ligament or meniscal injury to the index joint requiring at least one week of non weight bearing (minor ligamentous injury prior to 6 months is not an exclusion).
* Poor health that would impair compliance or assessment such as shortness of breath with exertion
* Neurological disease including vestibular dysfunction, or impaired vision
* Patient has a history of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient.
* Is unable to understand and complete the study questionnaires including visual analog scale (VAS) responses.
* Is unable to understand the study procedures.
* Investigator feels the patient is otherwise inappropriate for the study. The patient is participating in another clinical trial that would interfere with participation in this study
* Investigator feels the patient is otherwise inappropriate for the study.
* The patient is participating in another clinical trial that would interfere with participation in this study

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meika Fang, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West LA
Locations (1):
- VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California, United States

REFERENCES:
- [Derived] Fang MA, Heiney C, Yentes JM, Harada ND, Masih S, Perell-Gerson KL. Effects of contralateral versus ipsilateral cane use on gait in people with knee osteoarthritis. PM R. 2015 Apr;7(4):400-6. doi: 10.1016/j.pmrj.2014.09.018. Epub 2014 Oct 8. PMID 25305371
- [Derived] Harada N, Fong S, Heiney C, Yentes JM, Perell-Gerson KL, Fang MA. Evaluation of two cane instruments in older adults with knee osteoarthritis. J Rehabil Res Dev. 2014;51(2):275-83. doi: 10.1682/JRRD.2013.06.0140. PMID 24933725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited 2005-2008from the outpatient clinics of the VA West Los Angeles Healthcare Center, an urban tertiary academic hospital.
Groups:
- Arm 1 - Control/Crossover: No cane first, then single point cane
- Arm 2 - Cane: Single point cane first, then continue with single point cane
Period: First Intervention - Eight Weeks
Arm/Group | Arm 1 - Control/Crossover | Arm 2 - Cane
Started | 26 | 27
Completed | 19 | 18
Not Completed | 7 | 9
Not completed — Lost to Follow-up | 7 | 9
Period: Second Intervention - All Use Canes 4 mo
Arm/Group | Arm 1 - Control/Crossover | Arm 2 - Cane
Started | 19 | 18
Completed | 18 | 17
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Baseline Characteristics All Subjects: Community-dwelling patients with unilateral knee pain on movement which they scored at >35 mm on a 100-mm visual analogue scale (VAS) for most days of the previous month. Other inclusion criteria included having a weight less than 300 pounds, no cane use for the past 30 days, fulfillment of the American College of Rheumatology criteria for knee OA , and radiographic Kellgren-Lawrence scale knee OA grade > 1. We excluded individuals who had knee trauma or surgery, including arthroscopic surgery, within the past six months, upper body weakness, injury or amputation to the lower extremity joints, symptomatic spine, hip, ankle, or foot disease that would interfere with assessment of the knee, poor health that would impair compliance or assessment such as shortness of breath with exertion, or neurological disease including vestibular dysfunction, or impaired vision.
Arm/Group | Baseline Characteristics All Subjects
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 44
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Peak Vertical Force on Affected Limb
Description: An in-shoe dynamic, pressure distribution system (Pedar-X System, Novel Electronics, Inc., St. Paul, MN) was utilized to measure the vertical ground reaction force at the baseline visit and at the end of the first intervention period (two months) gait evaluations for both the control arm and cane user arm. The control arm was not given a cane to use at home during the two month intervention period. Peak vertical force on the affected limb was measured in the laboratory setting when both control group and cane user group walked with and without a cane at baseline and at the end of the first intervention period (2 months).
Time Frame: Baseline and end of first intervention period (2 months)
Measure: Mean (Standard Deviation); unit: N/kg
Groups:
- Arm 1 - Waiting Control: Study participants with symptomatic knee OA underwent gait analysis while walking with and without a cane at baseline and at end of first intervention period (2 months). Participants not given a cane to use at home during the intervention period. They were given a cane to use for four months after the first intervention period
- Arm 2- Cane Users: Study participants with symptomatic knee OA underwent gait analysis while walking with and without a cane at baseline and at end of first intervention period (2 months). Participants given a cane to use at home during the first intervention period and then for four months after the first intervention period.
Arm/Group | Arm 1 - Waiting Control | Arm 2- Cane Users
Number analyzed (Participants) | 26 | 27
N/kg
  Baseline - no cane | 9.5 (1.2) | 8.5 (1.8)
  Baseline - with cane | 8.8 (1.8) | 7.5 (1.8)
  2 months - no cane | 9.1 (1.1) | 8.9 (1.2)
  2 months - with cane | 8.3 (1.0) | 8.0 (1.2)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 6 month period.
Groups:
- Arm 1: Intervention - no Cane for First 8 Weeks: No cane for first 8 weeks
- Arm 1 - Intervention - Crossover to Cane: Given single point cane to use for 4 months following 8 weeks without a cane
- Arm 2- Single Point Cane: single point cane for 8 weeks then single point cane for next 4 months
Arm/Group | Arm 1: Intervention - no Cane for First 8 Weeks | Arm 1 - Intervention - Crossover to Cane | Arm 2- Single Point Cane
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/27

LIMITATIONS AND CAVEATS:
Had high drop out rate leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes